CLINICAL TRIAL: NCT04292704
Title: The Role of Fractional CO2 Laser in Consolidation Treatment of Recurrent Vulvovaginal Candidiasis (RVVC) ：a Study Protocol for a Randomized Controlled Trial
Brief Title: A Protocol for the Role of Fractional CO2 Laser in Consolidation Treatment of Recurrent Vulvovaginal Candidiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Shanghai Pudong Decoding Life Institutes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2020-07-101
Record Dates: First submitted 2020-02-24; First posted 2020-03-03 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Vulvovaginal Candidiasis, Genital; Laser Therapy
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Clotrimazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser group (Experimental): Fractional CO2 laser therapy in consolidation treatment once a month for 3 months and treatment was prohibited during menstrual period.
  Interventions: Radiation: the fractional CO2 laser
- Clotrimazole group (Other): Clotrimazole tablets 500mg PV biw q3d in consolidation treatment once a month for 6 months and treatment was prohibited during the menstrual period.
  Interventions: Drug: Clotrimazole

INTERVENTIONS:
Radiation: the fractional CO2 laser — The fractional CO2 laser therapy mechine: the wavelength is 10.6 μ m, the output power is 40 w, the action time is 2000 μ s and the lattice spacing is 700 ~ 1000 μ m
  Arms: Laser group
Drug: Clotrimazole — Clotrimazole vaginal tablets
  Arms: Clotrimazole group

SUMMARY:
Background: Recurrent vulvovaginal candidiasis (RVVC) is a common obstinate vulvovaginal inflammation in gynecology. At present, the pathogenesis of RVVC is not clear. In recent years, it is emphasized that the changes of vaginal microecological environment play an important role in the occurrence and development of RVVC. The treatment of RVVC can be divided into intensive treatment and consolidation treatment. Currently, local antifungal treatment is the main treatment regimen. While it is difficult and had an insufficient effect on prevention from recurrence of clinical signs and the improvement of vaginal mycological status in long term. Besides, there is no mature consolidation treatment regimen at home and abroad. Through the current application of the fractional CO2 laser in the treatment of atrophic vaginitis, it is confirmed that local irradiation of the fractional CO2 laser on vulva and vagina can regenerate and repair mucosal tissue, enhance the function of vaginal epithelial cells, gradually restore the normal pH value of vagina, improve vaginal microecological environment, restore the proportion of vaginal flora and reduce the recurrence rate of RVVC. This trial aims to explore the efficacy of two consolidation therapy schemes: the fractional CO2 laser and traditional antifungal drugs.

Methods/Design: The ongoing study will include 200 RVVC patients who voluntarily joined the study and signed the informed consent form the Second Affiliated Hospital of WMU during December 2019 to March 2022. After patients were cured by transvaginal local drug intensive therapy, participants will be randomly divided into control group (n = 100) and experimental group (n = 100). The control group continue to receive a monthly course of vaginal local drug consolidation therapy for 6 months, while the experimental group will be given monthly local vaginal CO2 laser consolidation therapy for 3 months. The vaginal secretions samples of RVVC patients will be collected before intensive therapy, after intensive therapy and at the end of consolidation therapy, and the species abundance and structure of vaginal flora were detected and analyzed. In the same period, 5 healthy women of childbearing age were recruited as the normal control group and the volunteers do not take any treatment. The vaginal secretions samples of 5 volunteers will be collected when signing the informed consent to detect and analyze the species abundance and structure of vaginal flora.

The patients with RVVC will be followed up for 3, 6 and 12 months after the treatment and vaginal secretions samples will be collected for vaginal flora structure detection to compare the vaginal microecological environment. For recurrent patients, the investigators will carry out targeted treatment, and again collect vaginal secretions sample to detect and analyze the species abundance and structure of vaginal flora.

Objectives: The aim of this study is to compare the effects of fractional CO2 laser consolidation therapy and traditional antifungal consolidation therapy for RVVC, and assess the role of fractional CO2 laser in changes of vaginal microecological environment and recurrence rate of VVC after consolidation treatment.

DETAILED DESCRIPTION:
1. Study design and general procedures

200 RVVC patients will be selected according to the above eligibility criteria form the Second Affiliated Hospital of WMU during December 2019 to March 2022. Women will be informed about the study protocol, procedures, investigational product and potential risks of treatment. After 200 RVVC patients were cured (mycological cured) by traditional intensive antifungal drug treatment, they will be randomly divided into control group (n=100) and experimental group (n=100). The control group continued to receive one course of Clotrimazole vaginal tablets for consolidation therapy once a month for 6 months, and the experimental group will be given the fractional CO2 laser therapy once a month for 3 months. In the same period, 5 healthy women of childbearing age will be recruited as the normal control group, and the normal control group do not receive any treatments.

2.Treatment

2.1 Intensive treatment: Clotrimazole tablets 500mg PV biw Q3d, with or without injector, the tablets are placed deep in the vagina for 2 weeks.

2.2 Consolidation treatment

2.2.1 Control group: Clotrimazole tablets 500mg PV biw q3d in consolidation therapy, with or without injector, the tablets are placed deep in the vagina once a month for 6 months. Treatment is prohibited during the menstrual period.

2.2.2 Experimental group: The fractional CO2 laser therapeutic machine will be used with wavelength 10.6 μ m, output power 40 w, action time 2000 μ s, lattice spacing 700 ~ 1000 μ m, gradually retreated from the vagina to the vaginal orifice according to the 5mm distance, and irradiated the vagina at 360 °once a month for 3 consecutive months as a course of treatment. Treatment is prohibited during menstrual period.

3. Sample collection and detection

3.1 Collection: Vaginal secretion samples will be collected from patients with RVVC before and after intensive therapy, at the end of consolidation therapy, and at 3, 6 and 12 months after consolidation therapy. The vaginal secretions samples of 5 volunteers will be collected when signing the informed consent. After emptying the urine, the participants take the lithotomy position in the gynecological examination bed, fully exposed the vulva and perineum. The gynecologists expose the cervix with a disposable vaginal dilator, collect the vaginal posterior fornix secretion with two disposable vaginal aseptic cotton swabs. Then the investigators send one sample to the Second Affiliated Hospital of WMU for vaginal discharge laboratory examination, put another sample into the 1.5ml cryopreservation tube and seal it in a liquid nitrogen tank at -80 ℃. These samples will be submitted to Shanghai Pudong Decoding Life Institutes for vaginal flora structure detection within 3 months.

3.2 Vaginal discharge laboratory examination: The Second Affiliated Hospital of WMU will take up the laboratory examination, including vaginal cleanliness, pH value of vagina, vaginal microbiological conditions. The use of a microscope to examine vaginal secretions wet smears and staining smears to observe their cleanliness and the presence of special bacteria and cells to confirm vaginal cleanliness and vaginal microbiological conditions. Vaginal pH value will be determined by the precise pH test paper method.

4. Follow-up visit: The investigatorswill take follow-up visit with RVVC patients at 3,6 and 12 months after consolidation therapy, and vaginal secretions samples will be collected for fungal culture to compare the vaginal microecological environment, evaluate clinical cure rate and recurrences of infection. Besides, the investigators will carry out targeted treatment for recurrent patients and again collect vaginal secretions sample to detect and analyze the species abundance and structure of vaginal flora.

5.Data analysis: ①By comparing the vaginal microecological environment (vaginal cleanliness, pH value of vagina, vaginal microbiological conditions and vaginal flora structure) between the normal control group (n=5) and 200 RVVC patients before the intensive therapy, the investigators will verify the vaginal microecological environment of RVVC patients has changed, and find out the difference between healthy women and RVVC patients. ②By comparing the vaginal microecological environment between control group (n=100) and experimental group (n=100) in different period (before and after intensive therapy, at the end of consolidation therapy, and at 3, 6 and 12 months after consolidation therapy), the investigators will find out the change of vaginal microecological environment in all treatment and development stages of RVVC, verify whether the fractional CO2 laser could restore the normal pH value of vagina, improve vaginal microecological environment, restore the proportion of vaginal flora or not. ③By comparing the cure rate and recurrence rate of VVC between control group (n=100) and experimental group (n=100) at 3, 6 and 12 months after consolidation therapy, the investigators can draw which treatment effect is better between fractional CO2 laser consolidation therapy and traditional antifungal consolidation therapy for RVVC.

ELIGIBILITY:
200 RVVC patients will be eligible for the trial if they fulfil the following criterion:

1. women aged 18 to 60;
2. chief complaint: vulvar itching, burning pain, sexual intercourse pain and urine pain, leucorrhea increased, occurring 4 or more times a year;
3. gynecological examination: vulvar erythema, edema, often accompanied by scratches, vaginal mucosa red and swollen, the inside of the labia minor and vaginal mucosa with white lumps, curd or bean curd-like, red and swollen mucous membrane exposed after erasure;
4. laboratory examination: microscopic examination of vaginal secretions to find the spores or hyphae of Candida albicans;
5. sign the informed consent form voluntarily.

5 healthy volunteers as the normal control group will be eligible for the trial if they fulfil the following criterion:

1. women aged 18 to 60;
2. no clinical symptoms;
3. vaginal cleanliness grade Ⅰ ~ Ⅱ;
4. laboratory examination: Candida spores or hyphae were not found in vaginal secretions;
5. menstruation was normal;
6. voluntary informed consent was signed.

Exclusion criteria:

1. those who did not meet the above inclusion criteria;
2. those with autoimmune or immunodeficiency diseases;
3. those who received antibiotics or antifungal therapy (including systemic and topical);
4. and special drugs and foods within 1 month;
5. women during lactation and pregnancy;
6. patients with liver insufficiency, neutropenia, adrenocortical dysfunction and diabetes;
7. those who are mentally abnormal and can not cooperate normally;
8. those who are allergic to clotrimazole vaginal tablets or other imidazole drugs.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 205 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
The difference of vaginal cleanliness between the healthy volunteers and 200 RVVC patients | before the intensive therapy
  Compare the vaginal cleanliness between the normal control group (n=5) and 200 RVVC patients. The criteria of vaginal cleanliness were as follow: Grade I was mainly gram-positive rods (indicative of Lactobacillus spp.), a large number of vaginal epithelial cells, and no other bacteria observed with WBC 0~5/HP under microscopy. Grade II was some Lactobacillus spp. and vaginal epithelial cells, some pus cells, and other bacteria observed under microscopy with WBC 10~15/HP. Grade III was a small amount of Lactobacillus spp. and vaginal epithelial cells, a large number of pus cells and other bacteria observed under microscopy with WBC 15~30/HP. Grade IV was no Lactobacillus spp., but pus cells and other bacteria observed under microscopy with WBC more than 30/HP.
The difference of the pH value of vagina between the healthy volunteers and 200 RVVC patients | before the intensive therapy
  Compare the pH value of vagina between the normal control group (n=5) and 200 RVVC patients. Vaginal pH value will be determined by the precise pH test paper method. The paper should include a range of pH from 4.0 to above 5.0. The normal pH is 4.5 or less.
The difference of vaginal microbiological conditions between the healthy volunteers and 200 RVVC patients | before the intensive therapy
  Compare the vaginal microbiological conditions between the normal control group (n=5) and 200 RVVC patients. Fungi, trichomonas, Neisseria gonorrhoeae and other items. If there is, then marked on the results "+" (positive), no is "-" (negative). Normal: none.
The difference of vaginal flora structure between the healthy volunteers and 200 RVVC patients | before the intensive therapy
  Compare the difference of vaginal flora structure between the normal control group (n=5) and 200 RVVC patients. The structure will be showed by the percentage of specific species (precent).
The changes of vaginal cleanliness between control group and experimental group in different period | up to 25 months
  Compare the vaginal cleanliness between control group (n=100) and experimental group (n=100) in different period (before and after intensive therapy, at the end of consolidation therapy, and at 3, 6 and 12 months after consolidation therapy). The criteria of vaginal cleanliness were as follow: Grade I was mainly gram-positive rods (indicative of Lactobacillus spp.), a large number of vaginal epithelial cells, and no other bacteria observed with WBC 0~5/HP under microscopy. Grade II was some Lactobacillus spp. and vaginal epithelial cells, some pus cells, and other bacteria observed under microscopy with WBC 10~15/HP. Grade III was a small amount of Lactobacillus spp. and vaginal epithelial cells, a large number of pus cells and other bacteria observed under microscopy with WBC 15~30/HP. Grade IV was no Lactobacillus spp., but pus cells and other bacteria observed under microscopy with WBC more than 30/HP.
The changes of the pH value of vagina between control group and experimental group in different period | up to 25 months
  Compare the pH value of vagina between control group (n=100) and experimental group (n=100) in different period (before and after intensive therapy, at the end of consolidation therapy, and at 3, 6 and 12 months after consolidation therapy). Vaginal pH value will be determined by the precise pH test paper method. The paper should include a range of pH from 4.0 to above 5.0. The normal pH is 4.5 or less.
The changes of the vaginal microbiological conditions between control group and experimental group in different period. | up to 25 months
  Compare the vaginal microbiological conditions between control group (n=100) and experimental group (n=100) in different period (before and after intensive therapy, at the end of consolidation therapy, and at 3, 6 and 12 months after consolidation therapy). Fungi, trichomonas, Neisseria gonorrhoeae and other items. If there is, then marked on the results "+" (positive), no is "-" (negative). Normal: none.
The changes of vaginal flora structure between control group and experimental group in different period. | up to 25 months
  Compare the vaginal flora structure between control group (n=100) and experimental group (n=100) in different period (before and after intensive therapy, at the end of consolidation therapy, and at 3, 6 and 12 months after consolidation therapy). The structure will be showed by the percentage of specific species (precent).
Cure rate | up to 25 months
  The criteria of cure: no clinical symptoms; vaginal cleanliness in gradeⅠ ~ Ⅱ; no Candida spores or hyphae were found in vaginal secretions samples detection at 3, 6 and 12 months after consolidation therapy. The rate of cured number in control group and experimental group (precent).
Recurrence rate of VVC | up to 25 months
  The criteria of recurrence: cured at the end of consolidation therapy, during the follow-up visit at 3,6 and 12 months after consolidation therapy, recurrence of VVC. The rate of recurrenced number in control group and experimental group (precent).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China